CLINICAL TRIAL: NCT04930341
Title: The Effect of Self-Acupressure Application on Pain, Fatigue and Sleep Quality in Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, PhD., Assistant Prof, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2308
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cancer
Keywords: Self-Acupressur; Cancer patients; Pain; Fatigue; Sleep quality
MeSH Terms: conditions — Neoplasms; Pain; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Single (Participant) Self-Acupressure and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Acupressure (Experimental): Each application to the acupressure points (H17, L14, ST36, SP6) will be done in 2 minutes and right and left)
  Interventions: Other: Self-Acupressure
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Self-Acupressure — Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in order to ensure the continuation and balance of the energy in our body.
  Arms: Self-Acupressure

SUMMARY:
The aim of this study is to examine the effect of Self-Acupressure application on pain, fatigue and sleep quality in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
Self-Acupressur application will improve pain, fatigue and sleep quality in cancer patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* To have received at least one course of adjuvant chemotherapy before,
* Not having a psychiatric diagnosis,
* Being an early stage cancer patient
* To be able to communicate adequately
* Not having psychiatric problems
* Volunteering to participate in research

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line.
  In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Visual Analog Scale | 4. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line.
  In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
The Piper Fatigue Scale | 1. week
  The Piper Fatigue Scale is a 22-item, self-reported scale. A total score of fatigue was recorded.
The Piper Fatigue Scale | 4. week
  The Piper Fatigue Scale is a 22-item, self-reported scale. A total score of fatigue was recorded.
Pittsburgh Sleep Quality Index (PSQI) | 1. week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | 4. week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz ÖZER, PhD, Study Chair — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He Y, Guo X, May BH, Zhang AL, Liu Y, Lu C, Mao JJ, Xue CC, Zhang H. Clinical Evidence for Association of Acupuncture and Acupressure With Improved Cancer Pain: A Systematic Review and Meta-Analysis. JAMA Oncol. 2020 Feb 1;6(2):271-278. doi: 10.1001/jamaoncol.2019.5233. PMID 31855257
- [Result] Dogan N, Tasci S. The Effects of Acupressure on Quality of Life and Dyspnea in Lung Cancer: A Randomized, Controlled Trial. Altern Ther Health Med. 2020 Jan;26(1):49-56. PMID 31221935